CLINICAL TRIAL: NCT03609567
Title: Aromatherapy as Treatment for Nausea and Vomiting of Pregnancy
Brief Title: Aromatherapy as Treatment for n/v of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4782
Record Dates: First submitted 2018-07-10; First posted 2018-08-01 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2018-07

CONDITIONS: Pregnancy Emesis
MeSH Terms: interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy (Experimental): Aromatherapy using essential oils
  Interventions: Other: Aromatherapy
- Placebo (Placebo Comparator): Aromatherapy using odorless placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Aromatherapy — Aromatherapy using essential oils
  Arms: Aromatherapy
Other: Placebo — Aromatherapy using odorless placebo oil
  Arms: Placebo

SUMMARY:
A double-blinded randomized controlled trial comparing essential oil aromatherapy versus placebo for treatment of first trimester nausea and vomiting of pregnancy.

DETAILED DESCRIPTION:
This is a double-blinded randomized controlled trial investigating the utility of essential oils for aromatherapy, compared to placebo, for treatment of nausea and vomiting in the first trimester of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy at <14 weeks gestation
* English-speaking
* Baseline PUQE score >=6

Exclusion Criteria:

* Non-compliant with prenatal care or study procedures
* Hyperemesis gravidarum
* Allergies to perfumes, essential oils or cosmetics
* Abnormal sense of smell
* Known acute or chronic GI disease
* Asthma
* Use of prescription anti-emetics

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Mean difference in Pregnancy-Unique Quantification of Emesis (PUQE) score | First trimester of pregnancy
  PUQE score is a validated measure of nausea and vomiting in pregnancy. It is a reliable tool used to measure the severity of nausea and vomiting of pregnancy. It is a questionnaire that measures the number of times in 24 hours a patient wretches, vomits, or feels nauseous. The minimum score is 3, and the maximum is 15. Participants will have PUQE scores calculated at baseline (during enrollment in the first trimester of pregnancy, at whatever age they are at), and after one month of aromatherapy use with either essential oils or placebo, with the mean difference from baseline compared as primary outcome. The Time Frame for participation will be from enrollment until the end of the first trimester (13th week of pregnancy), which, depending on gestational age in weeks at enrollment, may be up to 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Zelig, Study Chair — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No